CLINICAL TRIAL: NCT04398017
Title: Randomized Trial Comparing the Use of MEOPA (Equimolar Mixture of Nitrogen Protoxide and Oxygen)-Coupled Hypnosis Versus MEOPA Standard Care of Pain and Anxiety During Transesophageal Echocardiography (TEE) in Conscious Patients.
Brief Title: MEOPA-coupled Hypnosis Versus MEOPA-standard Care in Transesophageal Echocardiography
Acronym: HYPNETO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The early termination is due to an impossibility to include new candidates due to the degraded functioning of the service in connection with a chronic paramedical decrease in the number of caregivers trained in hypnosis.
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7351
Record Dates: First submitted 2020-01-22; First posted 2020-05-21 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Cardiac Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard support (Active Comparator)
  Interventions: Procedure: Transesophageal echography
- Hypnosis (Experimental)
  Interventions: Procedure: Transesophageal echography

INTERVENTIONS:
Procedure: Transesophageal echography — Ultrasound examination of the heart using a soft tube. The extremity is inserted through the mouth and positioned in the esophagus behind the heart.

SUMMARY:
The primary purpose is to evaluate the impact of hypnosis coupled with MEOPA (Equimolar Mix-ture of Nitrogen Protoxide and Oxygen) on patient comfort when performing transoesophageal echocardiographies.

Further studies on the use of MEOPA alone or the technique of hypnosis alone in the context of an TEE, would not be innovative in any way in view of previous studies or already in progress.

However, service has led to perform TEEs several times by combining MEOPA and hypnosis. Doctors noted a clear reduction in induction time for hypnosis and satisfaction of the patient and operators. This association technique is very often used in pediatrics.

According to one study, it seems that MEOPA increases the threshold of suggestibility and imagination. However suggestion and imagination are two essential notions of the hypnotic technique. To date, doctors have not found any other studies combining MEOPA and hypnosis for adults patients in the context of TEE.

This leads to the following hypothesis: Is there a difference for the patient in terms of for the global management of pain and anxiety between an TEE performed under MEOPA with a standard support and TEE under MEOPA coupled with hypnosis with support standard?

Secondary purposes are:

1. Compare patients' feelings / opinions: patients who have benefited from hypnosis associated with MEOPA versus patients who have been treated with MEOPA alone.
2. Compare patient stress: patients who have benefited from hypnosis associated with MEOPA versus patients who have benefited from MEOPA alone.
3. Compare the operators' feelings / opinions: procedures that have been performed under hypno-analgesia and MEOPA versus standard procedures under MEOPA alone.
4. Failed the TEE procedure

ELIGIBILITY:
Inclusion Criteria:

* Patient (male or female) of full age without upper age limit
* Patient hospitalized on the site of the Nouvel Hôpital Civil - Strasbourg, with an indication of transesophageal echography with a diagnostic purpose of a cardiac pathology (transesophageal echography scheduled the day after or the very day of selection)
* Patient affiliated to a social security health insurance scheme
* Patient able to understand the objectives and risks related to the research and to give an informed consent dated and signed
* For a woman of childbearing age: negative blood pregnancy test (test performed by the service as part of the care or diagnostic and therapeutic needs related to the patient's hospitalization).

Exclusion Criteria:

* Patient with a contraindication to the use of MEOPA
* Patient with little or no understanding of French
* Patient with hearing problems that do not allow hypnosis to occur
* Patient with psychiatric disorders (schizophrenia, psychosis, melancholic depression, hysteria...)
* Disoriented patients
* Patient receiving the following treatments/management:

ophthalmic gas centrally acting drugs: opiates, benzodiazepines and other psychotropic drugs (potentiation of effects).

* Long-term anxiolytics
* Premedications for transesophageal echocardiography by analgesics, Benzodiazepine, hydroxizine, antiemetics and gastric prokinetics or gabapentinoïdes (gabapentin, pregabaline)
* Psychocorporal therapies or complementary therapies during the period of hospitalization (psychotherapy, meditation, acupuncture...)
* Patient in exclusion period (determined by a previous or ongoing study),
* Impossibility of giving the patient informed information (patient in an emergency situation, difficulties in understanding, etc.)
* Pregnancy or breastfeeding reported by the patient
* Patients under curatorship, guardianship, protection of justice
* If the patient has an VAPS >8/10, the transesophageal echocardiography procedure and therefore its inclusion in the research will be postponed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Concomitant Measure of Pain and Anxiety | Change from baseline Concomitant Measure of Pain and Anxiety at 10 minutes transesophageal echography
  Measurements are made according to self-evaluation scales

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Strasbourg - France, Strasbourg, France